CLINICAL TRIAL: NCT01303354
Title: Lumbar Transforaminal Epidural Dexamethasone: A Prospective, Randomized, Double-Blind Clinical Trial
Brief Title: Lumbar Transforaminal Epidural Dexamethasone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahadian, Farshad M., M.D. (Individual)
Collaborators: San Diego Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Farshad M. Ahadian, M.D., Clinical Professor of Anesthesiology, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UCSD IRB 080582
Record Dates: First submitted 2011-02-04; First posted 2011-02-24 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2011-02

CONDITIONS: Radicular; Neuropathic, Lumbar, Lumbosacral
Keywords: Epidural, Transforaminal, Steroid Injection, Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- DXM 4 mg (Experimental): Dexamethasone 4 mg
  Interventions: Procedure: Lumbar Transforaminal Epidural Steroid Injection
- DXM 8 mg (Experimental): Dexamethasone 8 mg
  Interventions: Procedure: Lumbar Transforaminal Epidural Steroid Injection
- DXM 12 mg (Experimental): Dexamethasone 12 mg
  Interventions: Procedure: Lumbar Transforaminal Epidural Steroid Injection

INTERVENTIONS:
Procedure: Lumbar Transforaminal Epidural Steroid Injection

SUMMARY:
The aim of this study is to assess the effectiveness and safety of dexamethasone for transforaminal epidural steroid injection. A secondary aim of this study is to obtain data on the lowest most effective dose of dexamethasone for this treatment and the effective duration of effect.

DETAILED DESCRIPTION:
Transforaminal epidural steroid injections (TFESI) have been demonstrated to be an effective treatment for radicular pain. Over the last decade, rare but serious complications have been reported following transforaminal epidural steroid injections (TFESI). Recent research indicates that certain types of corticosteroids containing microscopic particles may be responsible for these adverse events. Dexamethasone (DXM) is a non-particulate cortico-steroid that has not been implicated in these adverse events. However, there is inadequate evidence up to date to support the use of Dexamethasone (DXM) for transforaminal epidural steroid injections (TFESI). This study aims to bridge that gap.

ELIGIBILITY:
Inclusion Criteria:

* adults age 18 years and older, unilateral lumbar radicular pain, baseline distal radicular lower extremity pain VAS score ≥ 5/10, and prior favorable response to TFESI

Exclusion Criteria:

* pregnancy, infection, coagulopathy, uncontrolled diabetes mellitus, history of allergy to iodinated contrast medium and interventional therapies for pain within 90 days prior to study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Radicular Pain Visual Analogue Scale (VAS) Score change from baseline | Baseline, 4 weeks, 8 weeks, 12 weeks post injection
  Reduction of pain from baseline at each time point.

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI)- change from baseline | Baseline, 4 weeks, 8 weeks, 12 weeks post injection
  Improvement of disability level from baseline at each time point
Subject Global Impression of Change (SGIC) | 4 weeks, 8 weeks, 12 weeks
  Allows comparison of Subject Global Impression of Change (SGIC) between groups at each time point
Subject Global Satisfaction Scale (SGSS) | 4 weeks, 8 weeks, 12 weeks post injection
  Allows comparison of Subject Global Satisfaction Scale (SGSS) among groups at each time point
Number of Subjects with Adverse Events as a Measure of Safety and Tolerability | Day of and 1 week post injection
  Subjects were specifically assessed for the following adverse events on day-of and one-week post injection: allergic reaction, neurovascular events, pain on injection, paresthesias during the procedure or dysesthesias post procedure, dural puncture, headache, meningismus, neck pain, arm pain, worsening of back pain, worsening of leg pain, facial flusing, mania, insomnia, agitation, hypertension, hyperglycemia. They were also asked to report any other side-effects or complications.

CONTACTS AND LOCATIONS:
Overall Officials: Farshad M Ahadian, M.D., Principal Investigator — University of California, San Diego
Locations (2):
- United States (2):
  - University of California, San Diego - Center for Pain Medicine, La Jolla, California
  - San Diego VA Healthcare System, La Jolla, California

REFERENCES:
- [Derived] Ahadian FM, McGreevy K, Schulteis G. Lumbar transforaminal epidural dexamethasone: a prospective, randomized, double-blind, dose-response trial. Reg Anesth Pain Med. 2011 Nov-Dec;36(6):572-8. doi: 10.1097/AAP.0b013e318232e843. PMID 22005659